CLINICAL TRIAL: NCT07196904
Title: A Randomized Controlled Clinical Trial Evaluating the Effectiveness of Ultrasonic Device in Impacted Mandibular Third Molar Surgery: Assessment Through Clinical Indices and Salivary C-reactive Protein Levels
Brief Title: Ultrasonic vs Rotary Instruments in Impacted Mandibular Third Molar Surgery: Clinical and Salivary CRP Outcomes
Acronym: PiezoCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Huynh Thien An (Other)
Responsible Party: Sponsor-Investigator, Le Huynh Thien An, Lecturer, Department of Oral Surgery, Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Piezo-CRP-2025; 1428/ĐHYD-HĐĐĐ (Other: Institutional Review Board, University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Impacted Mandibular Third Molar; Pain; Swelling; Trismus; Inflammation
MeSH Terms: conditions — Pain; Trismus; Inflammation | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic Device (Piezosurgery) (Experimental): Surgical extraction of impacted mandibular third molars using an ultrasonic surgical device (piezosurgery). Clinical outcomes (pain, swelling, trismus) and salivary hsCRP levels will be assessed.
  Interventions: Device: Ultrasonic Device (Piezosurgery)
- Conventional Rotary Instruments (Active Comparator): Surgical extraction of impacted mandibular third molars using conventional rotary instruments. Clinical outcomes (pain, swelling, trismus) and salivary hsCRP levels will be assessed.
  Interventions: Device: Conventional rotary instruments

INTERVENTIONS:
Device: Ultrasonic Device (Piezosurgery) — Mandibular impacted third molar extraction performed with an ultrasonic surgical device. The piezosurgery device was used exclusively for the osteotomy (bone removal) stage, while conventional rotary instruments were still used for tooth sectioning when required. This selective approach aimed to evaluate whether piezosurgery could reduce surgical trauma compared to full rotary techniques.
  Arms: Ultrasonic Device (Piezosurgery)
Device: Conventional rotary instruments — Mandibular impacted third molar extraction performed entirely with conventional rotary instruments. Both bone removal and tooth sectioning were conducted using high-speed rotary instruments under continuous irrigation. This served as the control arm to compare with the ultrasonic-assisted technique.
  Arms: Conventional Rotary Instruments

SUMMARY:
In the surgical removal of impacted mandibular third molars, ultrasonic surgical devices (piezosurgery) have been introduced with the expectation of reducing postoperative complications such as swelling, pain, and trismus, compared with conventional rotary instruments. To objectively evaluate the postoperative inflammatory response, salivary high-sensitivity C-reactive protein (hsCRP), a reliable biomarker of acute inflammation, will also be measured.

This randomized controlled clinical trial is designed to compare the effectiveness of ultrasonic surgery and conventional rotary instruments in impacted mandibular third molar extraction. The study has two primary objectives:

* To compare clinical outcomes, including swelling, mouth opening limitation, and pain, on postoperative days 2 and 5 between the two surgical methods.
* To assess changes in salivary hsCRP levels by comparing preoperative baseline values with postoperative day 2 values, and to determine differences between the two surgical techniques.

A total of 22 patients indicated for bilateral impacted mandibular third molar extractions of similar difficulty will be enrolled. Each patient will undergo one extraction using ultrasonic surgery and the contralateral extraction using rotary instruments, in a randomized split-mouth design.

Pain and swelling will be assessed on postoperative days 2 and 5. Saliva samples will be collected preoperatively and on postoperative day 2 for hsCRP analysis using enzyme-linked immunosorbent assay (ELISA).

The hypothesis is that ultrasonic surgery will result in reduced pain, swelling, and limitation of mouth opening, as well as lower salivary hsCRP levels, compared with conventional rotary instruments. Findings from this study may provide scientific evidence supporting the use of ultrasonic devices to improve patient outcomes and may highlight the role of salivary hsCRP as a non-invasive biomarker for monitoring inflammation after oral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA Physical Status index ≤ 2), aged 18-35 years.
* Patients presenting with bilateral impacted mandibular third molars of comparable difficulty, with the angulation difference between the two teeth not exceeding 15 degrees, as assessed according to the Pell and Gregory classification on panoramic radiographs.
* Patients who agree to participate in the study after being fully informed about the objectives and requirements.

Exclusion Criteria:

* Patients with acute systemic or oral infection at the surgical sites.
* Patients with clinical evidence of tumors or cystic lesions, or radiolucent lesions larger than 3 mm on radiographs at the mandibular third molar site.
* Patients with a history of antibiotic or anti-inflammatory drug use within 3 weeks prior to study participation.
* Patients with psychiatric disorders, motor dysfunction, or trauma in the maxillofacial region.
* Patients with systemic diseases or medication use that reduces salivary secretion, such as Sjögren's syndrome or prior head and neck radiotherapy.
* Pregnant or breastfeeding women.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Salivary hsCRP concentration | Preoperative (baseline) and day 2 after surgery
  High-sensitivity C-reactive protein (hsCRP) levels in saliva measured by ELISA assay. Baseline value before surgery will be compared with postoperative Day 2 levels to assess inflammatory response between groups.

SECONDARY OUTCOMES:
Postoperative pain | Day 2 and Day 5 post-surgery.
  Change in patient-reported pain intensity using a 10-point Visual Analog Scale (VAS), range 0-10, 0 = no pain, 10 = worst imaginable pain).
Postoperative swelling | Day 2 and Day 5 post-surgery
  Change in extraoral facial dimensions measured at specific anatomical landmarks
Mouth opening (trismus) | Day 2 and Day 5 post-surgery
  Change in maximum interincisal distance (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Faculty of Dentistry, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No